CLINICAL TRIAL: NCT02247700
Title: An Observational Cohort Study of Distribution of Ventilation in Infants and Children Requiring Mechanical Ventilation by Electrical Impedance Tomography
Brief Title: Observational Cohort Study of Distribution of Ventilation in Pediatrics Requiring Mechanical Ventilation by Electrical Impedance Tomography
Acronym: EIT
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Draeger Medical, Inc (Industry)
Responsible Party: Principal Investigator, Brian Walsh, Research Coordinator, Boston Children's Hospital
Other Study IDs: IRB-P00013295
Record Dates: First submitted 2014-07-02; First posted 2014-09-25 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Respiratory Failure; Acute Respiratory Distress Syndrome; Acute Lung Injury
Keywords: Pediatrics; ARDS; ARF; ALI; Respiratory; Mechanical ventilation; Ventilation; Noninvasive monitoring; electrical impedance tomography; EIT
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome; Acute Lung Injury; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mechanical Ventilation: Infants and Children requiring mechanical ventilation

SUMMARY:
Respiratory disorders are the leading cause of respiratory failure in children. Thousands of children are admitted to a pediatric intensive care unit each year and placed on mechanical ventilators. Despite over 40 years since the first pediatric-specific ventilator was designed, there has been no specific cardiopulmonary directed therapy that has proven superior. While mechanical ventilation is generally lifesaving, it can be associated with adverse events. There is evidence building to suggest that adopting a lung protective ventilation strategy by the avoidance of lung over-distension and collapse reduces death. Therefore, timely discovery of these two lung conditions is extremely important in order to mitigate the effects associated with positive pressure mechanical ventilation. The investigators research team has extensive research experience with a non-invasive and radiation free medical device called electrical impendence tomography (EIT). EIT is intended to generate regional information of changes in ventilation. Meaning it can detect this collapse and overdistension. This additional source of information could help fine tune the mechanical ventilator. A baseline of understanding of how often this occurs in the patients the investigators serve is required. Therefore the investigators propose an EIT observation study in their pediatric ICU patient population.

DETAILED DESCRIPTION:
A. Specific Aims/Objectives Specific Aim 1: To determine regional compliance and distribution of ventilation in a cohort of children requiring mechanical ventilation. Hypothesis - Abnormal distribution of ventilation will be discovered in all patients.

Specific Aim 2: To determine changes in regional distribution of ventilation over the course of mechanical ventilation therapy. Hypothesis - Distribution of regional ventilation will change significantly as the patient's lung function improves and as they progress towards liberation from mechanical ventilation.

Specific Aim 3: To compare previously developed EIT guided ventilation algorithms by BCH research team with medical team decisions regarding mechanical ventilation. Hypothesis - EIT guided ventilation algorithms will identify changes to minimize atelectasis and overdistension sooner than clinical team decisions.

B. Background and Significance Clinical decisions regarding the mechanical ventilator rely heavily on clinical judgment typically based on intermittent and subjective assessments of relevant physiologic parameters which only reflect global lung function and without consideration for regional distribution of ventilation. Until recently there has not been a way to determine regional distribution of ventilation without exposing a patient to radiation in the form of a chest radiograph (CXR) or computer aided tomography (CT). CT and CXR provide regionally specific information but only as a snapshot in time. Determining how different regions of the lung respond to therapeutic interventions over time is challenging. However, our research team has extensive research experience with a non-invasive and radiation free medical imaging technology called electrical impendence tomography (EIT). EIT provides regional information of changes in ventilation. This additional source of information could help optimize mechanical ventilation by providing bedside clinicians with continuous decision support as the EIT data may be utilized to alert when regional collapse or over-distension is detected. However, there is little data describing changes in distribution of ventilation over time or as the patient's condition changes.

Electrical Impedance Tomography (EIT) Barber and Brown introduced electrical impedance tomography to the medical community in the early 1980s. From there a wide spectrum of applications in medicine ranging from gastric emptying, brain function, breast imaging, to lung function have been explored. It is our belief that the most valuable benefit of EIT is in the monitoring of regional lung function in critically ill patients. Early EIT devices fell susceptible to poor sensitivity and signal interference in the clinical setting. After years and a renewed interest from a few commercial companies interested in ventilation technology, many of these shortcomings have been resolved. As with any new modality, EIT and its clinical utility and application need to be methodically explored; therefore we propose this IRB protocol to take us a step closer on this journey to develop a clinically useful tool9.

Electrical impedance tomography capitalizes on changes in electrical impendence between air-filled versus tissue or fluid-filled spaces in order to characterize and quantify regional distribution of lung volume at the bedside. This technology has been validated in animal10 and human11, 12 studies. The technology utilizes a series of 16 electrodes placed across the patient's chest. As small currents, which are undetectable to the subject, are passed between the electrodes, impedance is measured between and amongst the series. Through a complex interrogation and manipulation of these impedance values, a two-dimensional image is formed, and has been shown to correlate with clinical and radiographic changes in patients.11 The ability to estimate lung volume and regional distribution of gas non-invasively and in real time may give us insight as to what mode of ventilation or setting is more effective in optimizing positive pressure ventilation.

We have chosen to partner with Draeger Medical (Lubeck, Germany) through a CTA to explore the use of their commercially available product in Europe (not FDA cleared), through European Directive 93/42/EEC (medical devices) and meets the EN ISO 9001 and EN ISO 13485 requirements. Boston Children's Hospital has extensive experience with their prototype system that led to the final product named PulmoVista 500. The PulmoVista 500 uses 16 electrodes to measure the voltages utilized for image reconstruction. Mathematical simulations based on this electrode arrangement demonstrate a spatial resolution of 15% of the thoracic diameter; however the resolution decreases to 20% towards the center of the body. While CT scanners typically provide images consisting of 512 x 512 or higher pixels, EIT images from the PulmoVista 500 only consist of 32 x 32 pixels, which are 256 times less pixels when compared to CT images9. However, our team intends to use EIT at the bedside and within the ICU environment to guide ventilation therapy in the future rather than be a high-resolution diagnostic tool such as CT or MRI. Our intent is not to replace CT or MRI imaging of the lung, but develop a bedside tool to guide ventilation in the future that can be applied continuously and with very few risks. The characterization of a cohort of critically ill mechanically ventilated children, as proposed in this protocol represents an important step towards clinical utility of EIT.

C. Preliminary Studies Current strategies to provide lung protective ventilation rely on avoiding conditions associated with lung injury. There is growing interest in development of individualized mechanical ventilation treatment plans. The use of EIT has been demonstrated to be an accurate method of monitoring regional lung volume changes in animals and humans.10, 13, 14 While radiological and EIT images both provide information about the regional distribution of air in the lungs the image characteristics provided by these modalities are quite different. Radiological images of the lung provide information on the air content and reflect, depending on the moment the images were taken, the endinspiratory, the end-expiratory status or a lung condition somewhere in between. EIT images reflect the lung function, not the lung itself, which means EIT displays ventilated lung regions rather than morphological or anatomical structures of the lung.9 Nonetheless, the regional information contained in EIT and CT images is closely related to each other when pathological conditions such as pleural effusion or atelectasis lead to non-aerated and non-ventilated lung regions. While CT images display lungs regions with trapped air (e.g. pneumothorax) in black because of the large air content, EIT also displays those regions in black because they are not ventilated.15, 16 Conversely a CT image may indicate a region of consolidated lung tissue in a white color because of the high fluid content, while this region might be displayed in the EIT image in black or dark blue color, if this region is not or only partially ventilated.17 EIT has been proven in animal models and human case reports to be accurate determinant of pneumothoraces.15, 18, 19 More recently, EIT-derived parameters have been used to differentiate atelectatic, overdistened, and adequately recruited lung in different lung regions by a number of investigators.10, 20-28 Despite the ability of EIT to monitor regional lung behavior, the use of EIT derived indices has not been shown to improve outcomes in animals or humans with acute lung injury until last year when Drs. Wolf, Arnold and colleagues developed an EIT guided mechanical ventilation strategy that demonstrated promise in an animal model.29 Through this translational model they were able to demonstrate that EIT guided ventilation was superior to a national and standardized ventilation protocol called Acute Respiratory Distress Syndrome Network (ARDSNet) Ventilator Protocol.30-33 The goal of this study is to survey regional distribution in pediatric patients who require mechanical ventilation therapy.

D. Design and Methods (1) Study Design In a prospective observational trial we will objectively measure regional compliance and distribution of ventilation by EIT in patients who require mechanical ventilation.

(3) Description of Study Treatments or Exposures/Predictors Following attending approval and informed consent, patients who meet inclusion criteria and none of the exclusion criteria will (1) transition to the exact same setting on the FDA approved Draeger V500 ventilator. (2) A clinical assessment by the responsible respiratory therapist and nurse will be conducted to ensure the transitioned settings are appropriate and according to the standard of practice. (3) The PulmoVista 500 EIT device will be set-up and safety checked according to provided training and operating manual. (4) The provided electrode system will be placed around the patient's chest as in figure 2. (5) The EIT system will be connected to the electrodes array and the V500 ventilator. (6) Once signal quality is determined to be appropriate, a recording will be performed and saved securely. (7) The EIT belt and device will be removed and returned to storage and the V500 ventilator will remain on the patient for the ventilator course. The initial set-up and monitoring time commitment is approximately 1 hour. (8) Repeat recordings will be performed each morning for the first 5 days, then every other day if > 5 days of mechanical ventilation is required and within 2 hours following major interventions such as prone positioning, increasing or decrease of PEEP or MAP of 2 cmH2O or more, recruitment maneuvers, intubation (if on non-invasive ventilation), and prior to and following extubation. Follow-up monitoring events will be approximately 30 minutes. No set-up or monitoring session will be done without the approval of the bedside nurse and respiratory therapist.

Treatment exposures modification

Transition of the patient to the Draeger V500 Ventilator will not occur in the following situations:

1. Patients who are deemed too unstable by the research in collaboration with the medical team to transition to the V500, yet are stable enough to apply the EIT belt will be studied without the Draeger V500 ventilator. Manual recording of the ventilator settings and measurements will be conducted instead.
2. Patients enrolled who are receiving non-invasive ventilation. (5) Data Collection Methods, Assessments, Interventions and Schedule (what assessments performed, how often) Data will be collected from several sources. Initial evaluation will be performed within 48 hours of initiation of mechanical ventilation. Vital signs, latest blood gas, CXR report, ventilator settings, pulmonary mechanic and EIT images will be recorded. Vital signs will be gathered from T3. Blood gas will be captured from Powerchart. Pulmonary mechanics and EIT images will be obtained from the PulmoVista 500 system. The PulmoVista will obtain the ventilator settings and pulmonary mechanics via a connection to the Draeger V500 ventilator. A manual flowsheet (paper) of findings will be recorded and compared to the electronic files. Once verified, the manual flowsheet will be properly disposed.

The Pulmovista 500 system trends not only regional distribution of ventilation, but clinically useful and currently recorded information such as dynamic compliance, resistance, and ventilator settings. While the research team will not guide ventilation at this time from EIT images/data, the trending data summarized daily maybe useful. Parents will not be excluded from see the images if they desire. However, no data will be shared unless requested by the team. EIT images or data will not be used for routine clinical care or interventions, unless there is safety concern in which the team will be immediately notified and asked to clinically assess. Please see Risk/Benefit section of the online CHeRP protocol.

(6) Study Timeline (as applicable)

1. Initial set-up and recording will conducted as soon as possible following initiation of mechanical ventilation. Total set-up and recording is anticipated to take 1 hour.
2. Routine subsequent recordings will be conducted every morning for the first 5 days of mechanical ventilation; then every other day until liberation.
3. Interventional recordings will be conducted within 2 hours following changes of 2 cmH2O or more in PEEP or MAP, prone positioning, intubation, extubation, or modes of ventilation (inclusive of ECMO or HFV).

E. Adverse Event Criteria and Reporting Procedures The following complications will be monitored for during the imagining process which include study timelines 1-3 above and major complications will be immediately reported to the IRB. Minor events include: skin irritation that continues for > than 1 hour after the belt is removed, increase in respiratory rate by > 20%, temporal hypoventilation determined by an increase in ETCO2 by 10 mmHg, temporal increase in FIO2 of > 0.3, and temporal hypoxia determined by an desaturation (<88%) for greater than 1 minute. Minor events that occur more than 3 times will be reported to the IRB with a plan of action of how to avoid.

Major events that will halt the study and be immediately reported to the IRB are:

* Desaturation < 80% (continuously monitored by pulse oximetry) for longer than 1 minute.
* Bradycardia < 60 BPM
* Decrease in lung compliance determined to be associated with the belt. All adverse events will be reviewed by the entire research team weekly and a detailed case report will be developed. If major or minor events occurring more than 3 times, the study will not continue until the research team and IRB feel as though it is safe to continue.

F. Data Management Methods Upon entry, each patient will be assigned a number unique and unlinked from their medical record for the purpose of patient tracking. This number will be entered into a privately owned BCH, password protected research database (RedCap) accessible only by BCH study personnel.

A spreadsheet will be kept at the bedside during the data collection periods for each data point to be entered manually. This spreadsheet will be destroyed once the electric and manual data have been verified.

G. Quality Control Method Quality of the transfer of data will be ensured by a second investigator, who will confirm the manual and electronic data. RedCap and SPSS software will be used to help analyze the data and ensuring data integrity by establishing alerts for non-filled fields as well as unexpected or possibly misentered results.

H. Data Analysis Plan EIT data: The lung imaging system is the Dräger PulmoVista 500 (Dräger Medical, Lübeck, Germany). Sixteen coplanar electrodes will be placed equidistantly around the thorax at the level of the parasternal sixth intercostal space. The reference electrode will be placed on the right side of the abdomen near the waistline. Electrodes #1 and #16 are symmetrically placed to the left and the right of the sternum, respectively, so that electrodes #8 and #9 straddled the spinal column. This configuration leads to transverse images in the radiological convention, caudal to cranial, similar to a cat scan. Lung image reconstruction will be done according to the Graz consensus for electrical impedance tomography (GREIT)34 using the Electrical Impedance and Diffuse Optical Reconstruction Software.35 Each subjects' data will be filtered and images will be reconstructed using the aforementioned open source software platform. Each reconstructed lung image will then be segmented in to regions of interest and changes in impedance for each region will be transcribed. The procedure will be repeated for each of the individual subjects EIT recordings. Furthermore, we will employ, in an observational manner only, an algorithm which was developed by the current research group in order to identify when changes in lung mechanics are likely to reflect overdistention or collapse of lung.20 These discrete points, and the mechanical ventilator settings upon which they were collected will be transcribed and compared to the standard of care per unit practice. Impedance changes indicate how open or closed the lung is. This approach has been previously described in detail by our research group.20 I. Statistical Power and Sample Considerations Age Categories

1- < 6 months 6 months - < 1 year 1-7 years 8-14 years > 14 years This is a pilot observational study of mechanically ventilated children within our pediatric ICUs. We have proposed a target of 50 patients within two years. We anticipate a 10% dropout rate. Our goal would be to obtain 5-7 patients for each age category below. Since our experience and the preliminary data within this field is in severe lung injury and the fact that we wish to explore a heterogeneous mechanically ventilated patients, we have not been able to accurately determine a sample size and have therefore determined this to be a pilot study. Preference will be given to low volume lung disease patients such as but not limited to ARDS, CDH, hypoxic respiratory failure, patients transferred for possible ECMO, and asthmatics.

J. Study Organization Single institution pilot study.

ELIGIBILITY:
Inclusion Criteria:

* All patients who require mechanical ventilatory assistance. This includes invasive and noninvasive ventilation.
* Ages 1 day (full term defined as > 37 wks GA) to 17 years of age.

Exclusion Criteria:

* Patients with unstable spinal injuries or diseases
* Body mass index > 50
* Active implant such as pacemaker, ICD, or diaphragm pacer
* Patient who is having cardiac arrhythmias
* Skin integrity issues in the area that the belt / electrodes will be placed, such as ulcers or open wounds
* Dressings or chest tubes that prohibit the placement of electrodes in the proper plain.
* Open chest
* Flail chest within the regional plain of the belt / electrodes
* If the medical team feels that the patient is not appropriate to enroll in the study based on medical, social or emotional concerns
* If the patient is too unstable to position the belt / electrodes and/or transition to the Draeger ventilator
* Patient has been supported on mechanical ventilation for longer than 48 hours prior to enrollment
* Post-operative spinal fusion patients

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In a prospective observational trial we will objectively measure regional distribution of ventilation by EIT in patients who require mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2018-11-04 (Actual); Study Completion 2018-11-04 (Actual)

PRIMARY OUTCOMES:
Distribution of Ventilation | Every 24 hours or after PEEP changes
  Distribution of ventilation as determined by changes in impedence in layers or quarters.

SECONDARY OUTCOMES:
Distribution of Ventilation Changes Over Time | Every 24 hours for the duration of mechanical ventilation
  Changes if the distribution pattern over time

OTHER OUTCOMES:
EIT Guided Ventilation Algorithms | Images pre change in PEEP compared to post change
  Comparision of distribution of ventilation algorithms

CONTACTS AND LOCATIONS:
Overall Officials: Brian K Walsh, PhD, RRT, Principal Investigator — Boston Children's Hospital; John H Arnold, MD, Study Director — Boston Children's Hospital; Craig Smallwood, BS, RRT, Principal Investigator — Boston Children's Hospital; Jordan Rettig, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States